CLINICAL TRIAL: NCT03538262
Title: Tele-health Outcomes as Digital Biomarkers of Parkinson's Disease Progression During Extended Follow up of STEADY-PD3 and SURE-PD3 Trial Participants
Brief Title: Assessing Tele-Health Outcomes in Multiyear Extensions of PD Trials
Acronym: AT-HOME PD
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Northwestern University (Other); Sage Bionetworks (Other); University of Rochester (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Michael J. Fox Foundation for Parkinson's Research (Other); The Parkinson Study Group (Network)
Responsible Party: Principal Investigator, Michael Alan Schwarzschild, Professor of Neurology, Massachusetts General Hospital
Other Study IDs: AHPD-U01NS107009; U01NS090259-01A1 (NIH); U01NS080818-01A1 (NIH); U01NS080840-01A1 (NIH)
Record Dates: First submitted 2018-04-16; First posted 2018-05-29 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
Keywords: SURE-PD3; STEADY-PD III; Parkinson disease; PD; Parkinson Study Group (PSG); Telemedicine; Smartphone; Disease progression; Televisits; Patient-reported outcomes
MeSH Terms: conditions — Parkinson Disease; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- former phase 3 PD trial participants: The AT-HOME PD cohort enrolled upon completion of STEADY-PD3 or during completion of SURE-PD3; enrolling 2 to 6 years after diagnosis, and on standard dopaminergic therapy for 0 to 3 years. Former STEADY-PD3 participants had been randomized (1:1) to 3 years of isradipine or placebo treatment; SURE-PD3 participants had been randomized (1:1) to 2 years of inosine or placebo treatment.

SUMMARY:
An observational study to characterize and compare long-term clinical outcomes data collected remotely through periodic tele-visits, interactive smartphone app sessions, and web-based surveys in individuals with Parkinson's Disease (PD) who have completed the interventional phases of the STEADY-PD3 and SURE-PD3 clinical trials.

DETAILED DESCRIPTION:
Telemedicine and smartphone-based remote sensor assessments represent particularly promising opportunities to streamline study conduct, reduce participant burden, and allow for the collection of data beyond the usual episodic, in-clinic assessments. Demonstrating the utility of these relatively inexpensive accessible platforms for the measurement of PD progression would also establish the infrastructure for long-term follow up of participants after completion of interventional studies.

STEADY-PD3 (a.k.a. STEADY-PD III) and SURE-PD3 were both designed as phase 3 trials of potential disease-modifying interventions in PD. In both studies, de novo PD participants were randomized in 1:1 allocation to active therapy versus placebo with longitudinal follow up for three and two years, respectively. Both studies include collection of DNA and plasma samples, which along with rigorously collected clinical data will become part of the Parkinson's Disease Biomarker Program (PDBP), providing valuable resources for biomarker development. Long-term observation of participants from these two trials, together comprising ~600 early PD subjects, is invaluable not only in characterizing any persistent or delayed benefits of either randomized treatment but also in the development of tele-health outcomes to facilitate future interventional trials in PD and of neurotherapeutics more broadly.

Challenges of traditional long-term follow up of large cohorts are the high cost of in-clinic assessment, the high dropout rates and the need to maintain multi-site infrastructure. The objective of this study is to leverage modern technology to develop, pilot and implement a 100% virtual model for long-term follow up utilizing telemedicine and smartphone platforms for quantitative monitoring of clinician- and patient-reported outcomes (PROs). This cohort may also serve to test feasibility of new technology platforms as they become available.

ELIGIBILITY:
Inclusion Criteria:

1. Enrollment in STEADY-PD3 or SURE-PD3 studies
2. Prior consent to be contacted by the University of Rochester (UR) or if a participant from STEADY-PD III or SURE-PD3 studies directly contacts UR to request information about study participation
3. Internet-enabled device that will support participation in tele-visits
4. Have created or willing to create a Global Unique Identifier (GUID)
5. Willing and able to provide informed consent
6. English fluency
7. For participants opting to participate in the smartphone component, possession of a suitable smartphone (iPhone or Android) with adequate data plan and cellular network access/signal or wifi access

Exclusion Criteria:

1. Inability to carry out study activities as determined by study staff

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with early idiopathic PD enrolled in the STEADY-PD3 (a.k.a. STEADY-PD III; NCT02168842) and SURE-PD3 (NCT02642393) studies.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Schwarzschild, MD, PhD, Principal Investigator — Massachusetts General Hospital; Tanya Simuni, MD, Principal Investigator — Northwestern University; E. Ray Dorsey, MD, MBA, Principal Investigator — University of Rochester; Larsson Omberg, PhD, Principal Investigator — Sage Bionetworks
Locations (1):
- CHeT Telemedicine (Site 363), Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected across individual sites (University of Rochester for tele-visit data; Sage Bionetworks for smartphone data; MJFF-sponsored portal in the Laboratory of Neuroimaging (LONI) for FI PRO data). Data from all three sites will be aggregated in a centralized location using Synapse. Synapse is a cloud-based scientific data management and research collaboration platform designed and actively maintained by Sage Bionetworks (http://synapse.org) that is used to coordinate data across dozens of consortia and collaborations. All data will be aggregated following de-identification and coding by participant identification (ID)/Global Unique Identifier (GUID) within Synapse by Sage Bionetworks for analysis and for distribution to the Data Management Resource (DMR) of the Parkinson's Disease Biomarkers Program (PDBP) of the National Institutes for Health (NIH). The PDBP will ensure de-identified data sharing sharing with the broader research community per its public policies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: [per PDBP policy]
Access Criteria: [per PDBP policy]
URL: https://pdbp.ninds.nih.gov/policy

REFERENCES:
- See also: A nonprofit scientific network of North American centers for clinical studies of Parkinson disease — http://www.parkinson-study-group.org/
- See also: Parkinson's Disease BIomarkers Program (PDBP) of the National Institute of Neurological Disorders and Stroke (NINDS) — https://pdbp.ninds.nih.gov/
- See also: A nonprofit organization promoting open bioinformatics science and patient engagement in the research process; lead site for the smartphone app platform of AT-HOME PD. — http://sagebionetworks.org/
- See also: Center for Health + Technology (CHET) of the University of Rochester; lead site for the tele-visit platform of AT-HOME PD. — https://www.urmc.rochester.edu/health-technology.aspx
- See also: Fox Insight; online platform for the collection of patient-reported outcomes in AT-HOME PD. — https://foxinsight.michaeljfox.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Former Phase 3 PD Trial Participants
Started | 226
Completed | 203
Not Completed | 23

BASELINE CHARACTERISTICS:
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 220
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 215
  More than one race | 2
  Unknown or Not Reported | 0
Age at symptom onset [Mean (Standard Deviation); unit: years] | 59.4 (9.1)
Years from symptom onset to baseline [Mean (Standard Deviation); unit: years] | 5.30 (1.95)
Age at diagnosis [Mean (Standard Deviation); unit: years] | 60.9 (8.9)
Years from diagnosis to baseline [Mean (Standard Deviation); unit: years] | 3.82 (1.19)
Use of antiparkinsonian medications [Count of Participants; unit: Participants]
  No | 16
  Yes | 210
Use of levodopa [Count of Participants; unit: Participants]
  No | 62
  Yes | 164
MDS-UPDRS Part I [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorders Society Unified PD Rating Scale (MDS-UPDRS) Part I score comprises the responses to 13 questions on non-motor experiences of daily living. The first 6 responses are reported by the clinician (and constitute Part Ia), whereas the last 7 are patient-reported (and constitute Part Ib). The response to each question is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse disability. Part I scores may range from a minimum of 0 to a maximum of 52, with higher values meaning worse disability. Population: One participant did not complete MDS-UPDRS parts 1B and 2, which were administered as surveys via REDCap, at the baseline visit. Hence this participant does not have a baseline score for MDS-UPDRS Part I.
  units on a scale
    number analyzed (Participants) | 225
    (all) | 7.54 (4.84)
MDS-UPDRS Part Ia [Mean (Standard Deviation); unit: units on a scale] — Participants will be asked to complete (from home or other preferred environment) an hour-long Tele-visit that includes the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS), comprising MDS-UPDRS part 1a (i.e., the first six questions of part 1). The MDS-UPDRS is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse features. Part 1a scores may range from a minimum of 0 to a maximum of 24, with higher values meaning worse disability.
  units on a scale | 1.46 (2.10)
MDS-UPDRS Part Ib [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorders Society Unified PD Rating Scale (MDS-UPDRS) Part Ib is the patient-reported portion of Part I, and assesses non-motor experiences of daily living. The MDS-UPDRS is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse symptoms. Part Ib contains 7 questions, and its scores may range from a minimum of 0 to a maximum of 28, with higher values meaning worse symptoms. Population: One participant did not complete MDS-UPDRS parts 1B and 2, which were administered as surveys via REDCap, at the baseline visit.
  units on a scale
    number analyzed (Participants) | 225
    (all) | 6.08 (3.40)
MDS-UPDRS Part II [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorders Society Unified PD Rating Scale (MDS-UPDRS) Part II score comprises patient-reported responses to 13 questions on motor experiences of daily living. The response to each question is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse symptoms. Part II scores may range from a minimum of 0 to a maximum of 52, with higher values meaning worse symptoms. Population: One participant did not complete MDS-UPDRS parts 1B and 2, which were administered as surveys via REDCap, at the baseline visit.
  units on a scale
    number analyzed (Participants) | 225
    (all) | 8.60 (5.39)
MDS-UPDRS Part III [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (motor examination) is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse features. Total scores are calculated as simple sums of component items.
  units on a scale | 24.9 (11.5)
MDS-UPDRS Parts I-III Total Score [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse features. Total scores are calculated as simple sums of component items. Population: One participant did not complete MDS-UPDRS parts 1B and 2, which were administered as surveys via REDCap, at the baseline visit. Hence this participant does not have a baseline MDS-UPDRS Parts I-III total score.
  units on a scale
    number analyzed (Participants) | 225
    (all) | 41.0 (16.5)
MDS-UPDRS Part IV [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorders Society Unified PD Rating Scale (MDS-UPDRS) Part IV score comprises clinician-reported responses to 6 questions on motor complications of antiparkinsonian medication treatment. MDS-UPDRS Part IV is implemented only after a participant initiates symptomatic treatment with antiparkinsonian medication. The response to each question is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse symptoms. Part IV scores may range from a minimum of 0 to a maximum of 24, with higher values meaning worse symptoms. Population: 24 of the 226 participants are missing MDS-UPDRS Part 4 data at baseline.
  units on a scale
    number analyzed (Participants) | 202
    (all) | 2.42 (3.15)
Hoehn & Yahr [Mean (Standard Deviation); unit: units on a scale] — The Hoehn and Yahr Scale is an 6-level Parkinson's disease disability staging instrument. Its stages or values range from a minimum of 0 from to maximum of 5, with higher values meaning worse disability. Specifically, the values span from stage 0 meaning "no signs of disease" to stage 5 meaning "wheelchair bound or bedridden unless aided."
  units on a scale | 1.8 (0.4)
Schwab & England Activities of Daily Living (ADL) [Mean (Standard Deviation); unit: units on a scale] — The Schwab and England scale is a Site Investigator and subject assessment of the subject's level of independence. The subject will be scored on a percentage scale reflecting his/her ability to perform acts of daily living. Printed scores with associated descriptors range from 0% to 100% in increments of 5%, with higher percentages associated with more independence. A score of 0% implies "vegetative functions such as swallowing, bladder and bowel functions are not functioning; bedridden". A score of 100% implies "subject has full ability and is completely independent; essentially normal".
  units on a scale | 89.7 (8.3)
MoCA total score [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) assesses attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Points are awarded for the correct completion of MoCA tasks. Scores for each task are summed for a total score (range 0-30). Higher scores indicate greater cognitive capacity.
  units on a scale | 27.9 (2.0)
Clinician Global Impression - Severity [Count of Participants; unit: Participants] — The Clinician Global Impression (CGI) is an observer-rated scale that measures illness severity (CGIS). The CGIS is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through 7 (amongst the most severely ill patients).
  Participants
    1 = Normal, not at all incapacitated | 1
    2 = Borderline incapacitated | 60
    3 = Mildly incapacitated | 146
    4 = Moderately incapacitated | 19
Smartphone Tapping (Score) [Mean (Standard Deviation); unit: score on a scale] — The Smartphone Tapping Score is derived from a 30-second finger tapping task performed separately for each hand. The score ranges from 0 to 1 and higher scores are worse. Population: The analysis only includes subjects who consented to smartphone assessments.
  score on a scale
    number analyzed (Participants) | 178
    (all) | 0.627 (0.224)
Fox Insight MDS-UPDRS Part II Score [Mean (Standard Deviation); unit: score on a scale] — The Fox Insight MDS-UPDRS (Movement Disorders Society Unified PD Rating Scale) Part II score comprises patient-reported responses to 13 questions on motor experiences of daily living. Participants report their responses online through the Fox Insight web-based platform. The response to each question is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse symptoms. Part II scores may range from a minimum of 0 to a maximum of 52, with higher values meaning worse symptoms. Population: This is a self-completed assessment. Only assessments completed on schedule are reported.
  score on a scale
    number analyzed (Participants) | 93
    (all) | 7.978 (4.950)
Fox Insight PDQ-8 Score [Mean (Standard Deviation); unit: score on a scale] — The Fox Insight PDQ-8 (Parkinson's Disease Questionnaire, short-form 8 item version) is a self-administered questionnaire used to measure quality of life in persons with Parkinson's disease. The response to each question is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse symptoms. Scores range from a minimum of 0 to a maximum of 32, with a higher score indicating a poorer quality of life. Population: This is a self-completed assessment. Only assessments completed on schedule are reported.
  score on a scale
    number analyzed (Participants) | 120
    (all) | 2.927 (2.925)
Fox Insight EQ-5D Score [Mean (Standard Deviation); unit: score on a scale] — The Fox Insight EQ-5D (European Quality of life survey) is a standardized measure of health-related quality of life assessing 5 health dimensions (mobility, self-care, pain, usual activities, and physchological status), with 3 possible answers for each (1=no problem, 2=moderate problem, 3=severe problem). A derived summary index score is higher with better health-related quality of life. A maximum of 1 corresponds to the best quality of life, a score of 0 is intended to approximate a state equivalent to death, and values less than 1 correspond to a state worse than death. Population: This is a self-completed assessment. Only assessments completed on schedule are reported.
  score on a scale
    number analyzed (Participants) | 92
    (all) | 0.858 (0.132)
Fox Insight NMS-QUEST Score [Mean (Standard Deviation); unit: score on a scale] — The Non-motor Symptoms Questionnaire (NMS-QUEST) is a 30-question self-reported assessment. Each question is of a yes/no format with a score of 1 given to each "yes" answer, with total scores ranging from 0-30, with higher scores indicating a greater number of non-motor symptoms. Participants completed the assessment online in Fox Insight. Population: This is a self-completed assessment. Only assessments completed on schedule are reported.
  score on a scale
    number analyzed (Participants) | 120
    (all) | 6.950 (4.136)
Fox Insight REM (Rapid Eye Movement) Behavior Disorder Score [Mean (Standard Deviation); unit: score on a scale] — The Fox Insight Rapid Eye Movement Behavior Disorder (RBD) score is a patient-reported binary ("no" or "yes") response to a single question of whether they act out their dreams while asleep. Participants report their response online through the Fox Insight web-based platform. The score value is dichotomous (or missing) and ranges from 0 (no symptom) to 1 (yes response). Population: This is a self-completed assessment. Only assessments completed on schedule are reported.
  score on a scale
    number analyzed (Participants) | 75
    (all) | 0.373 (0.487)
Fox Insight PDAQ-15 Score [Mean (Standard Deviation); unit: score on a scale] — The Parkinson's Daily Activities Questionnaire -15 (PDAQ-15) is a 15-item measure of activities of daily living (ADL) that are impacted by cognitive impairment in participants with Parkinson's disease. The PDAQ-15 is derived from the original 50-item scale and is completed by the participant in Fox Insight. Scores range from 0 to 60, with higher scores indicating better function. Population: This is a self-completed assessment. Only assessments completed on schedule are reported.
  score on a scale
    number analyzed (Participants) | 90
    (all) | 55.444 (4.965)
Fox Insight GDS Score [Mean (Standard Deviation); unit: score on a scale] — The Geriatric Depression Scale (GDS) is a measure of depression completed by the participant online in Fox Insight. The scale has 30 yes/no questions, with each question having a maximum score of 1 and a total possible score ranging from 0 to 30. The higher the score, the greater the depression. Population: This is a self-completed assessment. Only assessments completed on schedule are reported.
  score on a scale
    number analyzed (Participants) | 78
    (all) | 1.830 (2.348)

OUTCOME MEASURES:

1. Primary Outcome: Change in Tele-visit Modified MDS-UPDRS Parts 1-3 (Total Score)
Description: Participants will be asked to complete (from home or other preferred environment) an hour-long Tele-visit that includes the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS), comprising MDS-UPDRS part 1a and (modified) part 3, as well as completion or confirmation of patient-reported component parts 1b and 2. The MDS-UPDRS is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse features. Parts I-III contain 59 total questions (13 in Part I, 13 in Part II, and 33 in Part III). Total scores are calculated as simple sums of component items with mean imputation by Part if no more than 1, 2, or 7 items are missing for Parts I through III, respectively. Total scores may range from 0 to 236, with 0 meaning no symptoms and 236 meaning worse symptoms.
Time Frame: Two years (0, 12, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 226
score on a scale
  BL to Month 12 | 2.197 [0.634 to 3.759]
  BL to Month 24 | 8.943 [6.920 to 10.966]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p = 0.006, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Test type: Other — Statistical analysis for BL to Month 24; p < 0.001, Mixed Models Analysis

2. Primary Outcome: Change in Tele-visit MDS-UPDRS Part 2 (Score)
Description: The Movement Disorders Society Unified PD Rating Scale (MDS-UPDRS) Part II score comprises patient-reported responses to 13 questions on motor experiences of daily living. The response to each question is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse symptoms. Part II scores may range from a minimum of 0 to a maximum of 52, with higher values meaning worse symptoms.
Time Frame: Two years (0, 12, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 226
score on a scale
  BL to Month 12 | 0.575 [0.134 to 1.017]
  BL to Month 24 | 1.550 [0.992 to 2.107]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p = 0.011, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 24; Test type: Other; p < 0.001, Mixed Models Analysis

3. Primary Outcome: Change in Smartphone Tapping (Score)
Description: The Smartphone Tapping Score is derived from a 30-second finger tapping task performed separately for each hand. The score ranges from 0 to 1 and higher scores are worse.
Time Frame: Two years (0, 3, 6, 9, 12 , 15, 18, 21, and 24 months)
Population: Only subjects who consented and enrolled in the smartphone assessments are included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 184
score on a scale
  BL to Month 3 | -0.051 [-0.088 to -0.014]
  BL to Month 6 | -0.088 [-0.122 to -0.053]
  BL to Month 9 | -0.057 [-0.096 to -0.019]
  BL to Month 12 | -0.078 [-0.108 to -0.049]
  BL to Month 15 | -0.106 [-0.138 to -0.075]
  BL to Month 18 | -0.116 [-0.149 to -0.082]
  BL to Month 21 | -0.114 [-0.150 to -0.077]
  BL to Month 24 | -0.139 [-0.175 to -0.102]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 3; Test type: Other; p = 0.007, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 6; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 9; Test type: Other; p = 0.004, Mixed Models Analysis
Statistical Analysis 4: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 5: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 15; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 6: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 18; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 7: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 21; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 8: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 24; Test type: Other; p < 0.001, Mixed Models Analysis

4. Primary Outcome: Change in Fox Insight MDS-UPDRS Part 2 (Score)
Description: The Fox Insight MDS-UPDRS (Movement Disorders Society Unified PD Rating Scale) Part II score comprises patient-reported responses to 13 questions on motor experiences of daily living. Participants report their responses online through the Fox Insight web-based platform. The response to each question is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse symptoms. Part II scores may range from a minimum of 0 to a maximum of 52, with higher values meaning worse symptoms.
Time Frame: Two years (0, 6, 12, 18, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 148
score on a scale
  BL to Month 6 | -0.002 [-0.837 to 0.833]
  BL to Month 12 | 1.027 [-0.017 to 2.070]
  BL to Month 18 | 1.367 [0.174 to 2.560]
  BL to Month 24 | 1.771 [0.522 to 3.020]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 6; Test type: Other; p = 0.996, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p = 0.054, Mixed Models Analysis
Statistical Analysis 3: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 18; Test type: Other; p = 0.025, Mixed Models Analysis
Statistical Analysis 4: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 24; Test type: Other; p = 0.006, Mixed Models Analysis

5. Secondary Outcome: Change in Tele-visit MDS-UPDRS Part 1a (Score)
Description: Participants will be asked to complete (from home or other preferred environment) an hour-long Tele-visit that includes the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS), comprising MDS-UPDRS part 1a (i.e., the first six questions of part 1). The MDS-UPDRS is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse features. Part 1a scores may range from a minimum of 0 to a maximum of 24, with higher values meaning worse disability.
Time Frame: Two years (0, 12, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 226
score on a scale
  BL to Month 12 | 0.189 [-0.066 to 0.445]
  BL to Month 24 | 0.313 [0.033 to 0.594]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p = 0.145, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 24; Test type: Other; p = 0.029, Mixed Models Analysis

6. Secondary Outcome: Change in Tele-visit MDS-UPDRS Part 1b (Score)
Description: The Movement Disorders Society Unified PD Rating Scale (MDS-UPDRS) Part Ib is the patient-reported portion of Part I, and assesses non-motor experiences of daily living. The MDS-UPDRS is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse symptoms. Part Ib contains 7 questions, and its scores may range from a minimum of 0 to a maximum of 28, with higher values meaning worse symptoms.
Time Frame: Two years (0, 12, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 226
score on a scale
  BL to Month 12 | 1.026 [0.667 to 1.384]
  BL to Month 24 | 1.238 [0.864 to 1.613]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p < .001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 24; Test type: Other; p < 0.001, Mixed Models Analysis

7. Secondary Outcome: Change in Tele-visit Modified MDS-UPDRS Part 3 (Score)
Description: Participants will be asked to complete (from home or other preferred environment) an hour-long Tele-visit that includes the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS), comprising MDS-UPDRS (modified) part 3. This measure omits 5 questions related to rigidity and 1 question related to postural instability, with a range from 0 to 108. The MDS-UPDRS is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse features.
Time Frame: Two years (0, 12, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 226
score on a scale
  BL to Month 12 | 0.457 [-0.572 to 1.486]
  BL to Month 24 | 4.617 [3.245 to 5.989]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p = 0.382, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 24; Test type: Other; p < 0.001, Mixed Models Analysis

8. Secondary Outcome: Change in Tele-visit Montreal Cognitive Assessment (MoCA; Score)
Description: The Montreal Cognitive Assessment (MoCA) assesses attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Points are awarded for the correct completion of MoCA tasks. Scores for each task are summed for a total score (range 0-30). Higher scores indicate greater cognitive capacity.
Time Frame: Two years (0, 12, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 226
score on a scale
  BL to Month 12 | -0.051 [-0.301 to 0.199]
  BL to Month 24 | 0.142 [-0.124 to 0.408]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Secondary analysis for BL to Month 12; Test type: Other; p = 0.688, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Secondary analysis for BL to Month 24; Test type: Other; p = 0.293, Mixed Models Analysis

9. Secondary Outcome: Change in Tele-visit Schwab and England (S&E; Score)
Description: The Schwab and England scale is a Site Investigator and subject assessment of the subject's level of independence. The subject will be scored on a percentage scale reflecting his/her ability to perform acts of daily living. Printed scores with associated descriptors range from 0% to 100% in increments of 5%, with higher percentages associated with more independence. A score of 0% implies "vegetative functions such as swallowing, bladder and bowel functions are not functioning; bedridden". A score of 100% implies "subject has full ability and is completely independent; essentially normal".
Time Frame: Two years (0, 12, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 226
score on a scale
  BL to Month 12 | -0.440 [-1.577 to 0.697]
  BL to Month 24 | -0.338 [-1.495 to 0.818]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p = 0.446, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 24; Test type: Other; p = 0.565, Mixed Models Analysis

10. Secondary Outcome: Change in Tele-visit Clinician Global Impression - Severity (CGIS; Score)
Description: The Clinician Global Impression (CGI) is an observer-rated scale that measures illness severity (CGIS). The CGIS is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through 7 (amongst the most severely ill patients).
Time Frame: Two years (0, 12, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 226
score on a scale
  BL to Month 12 | 0.103 [0.030 to 0.176]
  BL to Month 24 | 0.004 [-0.108 to 0.116]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p = 0.006, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 24; Test type: Other; p = 0.937, Mixed Models Analysis

11. Secondary Outcome: Change in Fox Insight Parkinson's Disease Questionnaire - 8 Item Version (PDQ-8; Score)
Description: The Fox Insight PDQ-8 (Parkinson's Disease Questionnaire, short-form 8 item version) is a self-administered questionnaire used to measure quality of life in persons with Parkinson's disease. The response to each question is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse symptoms. Scores range from a minimum of 0 to a maximum of 32, with a higher score indicating a poorer quality of life.
Time Frame: Two years (0, 3, 6, 9, 12, 15, 18, 21, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 154
score on a scale
  BL to Month 3 | 0.396 [0.016 to 0.775]
  BL to Month 6 | 0.637 [0.273 to 1.000]
  BL to Month 9 | 1.258 [0.849 to 1.667]
  BL to Month 12 | 1.113 [0.719 to 1.508]
  BL to Month 15 | 1.687 [1.208 to 2.166]
  BL to Month 18 | 1.543 [1.090 to 1.995]
  BL to Month 21 | 1.317 [0.894 to 1.740]
  BL to Month 24 | 1.744 [1.280 to 2.208]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 3; Test type: Other; p = 0.041, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 6; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 9; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 4: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 5: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 15; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 6: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 18; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 7: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 21; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 8: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 24; Test type: Other; p < 0.001, Mixed Models Analysis

12. Secondary Outcome: Change in Fox Insight EuroQol Five Dimensions Questionnaire (EQ-5D; Score)
Description: The Fox Insight EQ-5D (European Quality of life survey) is a standardized measure of health-related quality of life assessing five dimensions of health. It comprises five corresponding questions on mobility, self-care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem). A derived summary index score is higher with better health-related quality of life. A maximum of 1 corresponds to the best quality of life, whereas a score of 0 is intended to approximate a state equivalent to death, with values less than 1 corresponding to a state worse than death.
Time Frame: Two years (0, 6, 12, 18, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 146
score on a scale
  BL to Month 6 | -0.010 [-0.048 to 0.028]
  BL to Month 12 | -0.015 [-0.055 to 0.024]
  BL to Month 18 | 0.003 [-0.043 to 0.048]
  BL to Month 24 | -0.040 [-0.084 to 0.003]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 6; Test type: Other; p = 0.595, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p = 0.440, Mixed Models Analysis
Statistical Analysis 3: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 18; Test type: Other; p = 0.909, Mixed Models Analysis
Statistical Analysis 4: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 24; Test type: Other; p = 0.068, Mixed Models Analysis

13. Secondary Outcome: Change in Fox Insight Non-motor Symptoms Questionnaire (NMS-QUEST; Score)
Description: The Non-motor Symptoms Questionnaire (NMS-QUEST) is a 30-question self-reported assessment. Each question is of a yes/no format with a score of 1 given to each "yes" answer, with total scores ranging from 0-30, with higher scores indicating a greater number of non-motor symptoms. Participants completed the assessment online in Fox Insight.
Time Frame: Two years (0, 3, 6, 9, 12, 15, 18, 21, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 154
score on a scale
  BL to Month 3 | 0.447 [-0.043 to 0.938]
  BL to Month 6 | 1.062 [0.567 to 1.557]
  BL to Month 9 | 1.432 [0.914 to 1.950]
  BL to Month 12 | 1.323 [0.849 to 1.797]
  BL to Month 15 | 1.642 [1.122 to 2.163]
  BL to Month 18 | 1.720 [1.160 to 2.280]
  BL to Month 21 | 1.660 [1.092 to 2.227]
  BL to Month 24 | 2.046 [1.505 to 2.588]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 3; Test type: Other; p = 0.074, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 6; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 9; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 4: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 5: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 15; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 6: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 18; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 7: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 21; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 8: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 24; Test type: Other; p < 0.001, Mixed Models Analysis

14. Secondary Outcome: Change in Fox Insight REM (Rapid Eye Movement) Behavior Disorder (RBD; Score)
Description: The Fox Insight Rapid Eye Movement Behavior Disorder (RBD) score is a patient-reported binary ("no" or "yes") response to a single question of whether they act out their dreams while asleep. Participants report their response online through the Fox Insight web-based platform. The score value is dichotomous (or missing) and ranges from 0 (no symptom) to 1 (yes response).
Time Frame: Two years (0, 3, 6, 9, 12, 15, 18, 21, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 143
score on a scale
  BL to Month 3 | -0.125 [-0.318 to 0.068]
  BL to Month 6 | -0.008 [-0.128 to 0.111]
  BL to Month 9 | 0.020 [-0.177 to 0.217]
  BL to Month 12 | 0.088 [-0.124 to 0.300]
  BL to Month 15 | -0.117 [-0.327 to 0.094]
  BL to Month 18 | 0.148 [0.007 to 0.288]
  BL to Month 21 | 0.003 [-0.241 to 0.248]
  BL to Month 24 | 0.349 [0.081 to 0.616]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 3; Test type: Other; p = 0.200, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 6; Test type: Other; p = 0.888, Mixed Models Analysis
Statistical Analysis 3: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 9; Test type: Other; p = 0.837, Mixed Models Analysis
Statistical Analysis 4: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p = 0.394, Mixed Models Analysis
Statistical Analysis 5: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 15; Test type: Other; p = 0.268, Mixed Models Analysis
Statistical Analysis 6: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 18; Test type: Other; p = 0.039, Mixed Models Analysis
Statistical Analysis 7: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 21; Test type: Other; p = 0.979, Mixed Models Analysis
Statistical Analysis 8: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 24; Test type: Other; p = 0.014, Mixed Models Analysis

15. Secondary Outcome: Change in Fox Insight Parkinson's Daily Activities Questionnaire -15 (PDAQ-15; Score)
Description: The Parkinson's Daily Activities Questionnaire -15 (PDAQ-15) is a 15-item measure of activities of daily living (ADL) that are impacted by cognitive impairment in participants with Parkinson's disease. The PDAQ-15 is derived from the original 50-item scale and is completed by the participant in Fox Insight. Scores range from 0 to 60, with higher scores indicating better function.
Time Frame: Two years (0, 3, 9, 15, and 21 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 152
score on a scale
  BL to Month 3 | 0.611 [-0.514 to 1.735]
  BL to Month 9 | -0.798 [-2.218 to 0.621]
  BL to Month 15 | -0.400 [-1.769 to 0.970]
  BL to Month 21 | -1.618 [-3.105 to -0.130]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 3; Test type: Other; p = 0.285, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 9; Test type: Other; p = 0.267, Mixed Models Analysis
Statistical Analysis 3: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 15; Test type: Other; p = 0.564, Mixed Models Analysis
Statistical Analysis 4: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 21; Test type: Other; p = 0.034, Mixed Models Analysis

16. Secondary Outcome: Change in Fox Insight Geriatric Depression Scale (GDS; Score)
Description: The Geriatric Depression Scale (GDS) is a measure of depression completed by the participant online in Fox Insight. The scale has 30 yes/no questions, with each question having a maximum score of 1 and a total possible score ranging from 0 to 30. The higher the score, the greater the depression.
Time Frame: Two years (0, 12, and 24 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Former Phase 3 PD Trial Participants
Number analyzed (Participants) | 144
score on a scale
  BL to Month 12 | 0.401 [-0.581 to 1.382]
  BL to Month 24 | 0.855 [-0.330 to 2.040]
Statistical Analysis 1: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 12; Test type: Other; p = 0.409, Mixed Models Analysis
Statistical Analysis 2: Comparison: Former Phase 3 PD Trial Participants; Statistical analysis for BL to Month 0.149; Test type: Other; p = 0.149, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Former Phase 3 PD Trial Participants
All-Cause Mortality (participants affected / at risk) | 0/226
Serious Adverse Events (participants affected / at risk) | 0/226
Other Adverse Events (participants affected / at risk) | 1/226
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Former Phase 3 PD Trial Participants (N=226)
Fall (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
Per the study protocol, certain smartphone cognitive assessments were planned. However, smartphone cognitive assessments were not completed in this study due to the measures still being validated at the time of the study launch and being deployed too late to collect longitudinal data on the cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT03538262/Prot_SAP_000.pdf